CLINICAL TRIAL: NCT06578026
Title: Developing Resilience Skills and Social Competence in Youth in a School Setting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Catholic University of America (Other)
Responsible Party: Principal Investigator, Brendan Rich, Associate Professor, The Catholic University of America
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 16-057
Record Dates: First submitted 2024-08-24; First posted 2024-08-29 (Actual); Last update posted 2024-08-29 (Actual); Status verified 2024-08

CONDITIONS: Psychosocial Functioning
Keywords: resilience

STUDY DESIGN:
Intervention Model Description: randomized control trial
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment (Experimental): Received the Resilience Builder Program intervention
  Interventions: Behavioral: Resilience Builder Program
- Control (No Intervention): Did not receive the Resilience Builder Program

INTERVENTIONS:
Behavioral: Resilience Builder Program — The Resilience Builder Program® group therapy will meet for one class period once a week during the semester (12 sessions). The group aims to improve resilience skills: areas such as the ability to control emotions and behavior, social skills and interactions with peers, problem-solving skills, ability to be flexible in different situations, self-esteem, and optimistic thinking. The groups involve the group leader presenting a new topic and skill, the students discussing this topic and developing strategies associated with the skill, the students practicing the skill while getting feedback from the group leader, and a period focused on self-control strategies. A letter reviewing each session will be sent home to the parent/guardian each week. Also, each child will be asked to do an assignment between weekly sessions to help him/her practice new skills.
  Arms: Treatment

SUMMARY:
Our study aimed to answer the question: Can a resilience-based intervention improve the psychosocial and educational outcomes of students with psychosocial difficulties? We examined the effectiveness of a resilience-based group intervention, the Resilience Builder Program® (RBP), with students in low-SES school settings to determine if this treatment improves psychosocial and educational outcomes.

DETAILED DESCRIPTION:
Enhancing resilience is valuable to youth from economically marginalized communities given that they often face greater challenges and hardships than their peers from more affluent communities.

Efforts to increase resilience skills in these youth are hampered because they disproportionately encounter barriers in access to mental health interventions. Implementing school-based services may be optimal to address these inequalities. This project explores the effectiveness of a school-based group intervention (the Resilience Builder Program®) related to resilience and academic functioning in a sample of children from economically marginalized communities. Students (N = 169) with social-emotional difficulties were recruited from five elementary schools and randomly assigned to participate in the Resilience Builder Program® (RBP) immediately or following a semester delay. Participants, their parents, and teachers completed measures of resilience and academic functioning. Repeated-measures analysis of variance compares groups across time (pre-, post-intervention) on psychosocial and academic outcomes.

ELIGIBILITY:
Inclusion Criteria:

* psychosocial deficits

Exclusion Criteria:

* psychosis
* extreme aggression
* autism

Ages: 9 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 169 (Actual)
Dates: Start 2016-06-16 (Actual); Primary Completion 2020-03-13 (Actual); Study Completion 2020-03-13 (Actual)

PRIMARY OUTCOMES:
Resiliency scales for children and adolescent (RSCA) | 1 month
  self-report of child's resilience; score 0-100; higher scores = stronger resilience

SECONDARY OUTCOMES:
Behavior assessment system for children, 2nd edition (BASC) | 1 month
  parent, child, and teacher report across varied psychosocial subscales; score 0-100; scores vary based on subscale, higher scores can indicate greater impairment or better functioning

OTHER OUTCOMES:
Academic competence evaluation scales (ACES) | 1 month
  teacher report of student's academic engagement and motivation; score 0-100; higher scores = better functioning

CONTACTS AND LOCATIONS:
Locations (1):
- Montgomery County Public Schools, Rockville, Maryland, United States

IPD SHARING:
Plan to Share IPD: No
No plans to share with other researchers